CLINICAL TRIAL: NCT07304063
Title: Let's Talk: Overcoming Barriers to Uptake of Cascade Screening Through a Stakeholder-informed Online Intervention
Brief Title: Overcoming Barriers to Uptake of Cascade Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2516-AIM2; R21HG013417 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lynch Syndrome
Keywords: Screening; cascade screening
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Masking Description: 15 patients and 5 Genetic Counselor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic Counselor participants (Experimental): Participants who are practicing genetic counselor at a medical institution.
  Interventions: Behavioral: Let's Talk Genetics Providers
- Patient participants (Experimental): Participants who are with diagnosis of Lynch syndrome.
  Interventions: Behavioral: Let's Talk Patients

INTERVENTIONS:
Behavioral: Let's Talk Genetics Providers — Providers will complete a brief pre-intervention survey and a short training on the Let's Talk tool. They will then help recruit eligible patients from genetics clinics who need cascade screening for Lynch syndrome. After the intervention, providers will complete post-intervention surveys and interviews.
  Arms: Genetic Counselor participants
Behavioral: Let's Talk Patients — Patients will complete a brief pre-intervention survey and receive access to the online Let's Talk toolkit for two months. The toolkit addresses key barriers to cascade screening for Lynch syndrome by building knowledge, confidence, and communication skills through simple, evidence-based activities. After two months, patients will complete a post-intervention survey and participate in a qualitative interview.
  Arms: Patient participants

SUMMARY:
Lynch syndrome is a genetic condition that increases cancer risk. The public health impact of genetic testing for disease prevention hinges on cascade screening, which is the systematic identification and testing of blood relatives after a family member has been diagnosed with a genetic condition. Despite its importance in disease prevention, only half of first-degree relatives of individuals with Lynch syndrome undergo cascade screening. To address this gap, the study will pilot test an online version of Let's Talk, a novel intervention designed to support and promote cascade screening. This intervention tool is designed to support and encourage more family members to get screened. The purpose of this study aim is to assess the feasibility of the online Let's Talk tool in clinical use by examining implementation and effectiveness outcomes related to the use of the planning tool across three clinics at a large academic-affiliated medical center with patients (n=15) seen by one of five genetic counselors (n=5).

DETAILED DESCRIPTION:
The overall objective of this research study is to design an interactive online format for Let's Talk content, and pilot test Let's Talk to gain feasibility data for its clinical use among patients diagnosed with Lynch syndrome. The rationale for this study is that it has the potential to improve cascade screening uptake and could be adapted to other hereditary conditions in future work. The expected outcomes of this project will move the field forward in addressing barriers to cascade screening and will inform cascade screening for Lynch syndrome as well as for other conditions, such as hereditary breast and ovarian cancer syndrome and familial hypercholesterolemia.

Initially designed to support patients with Lynch Syndrome, Let's Talk is a theory-based intervention developed using a stakeholder engaged methodology that is responsive to reported barriers to cascade screening. Let's Talk was created in collaboration with patients and providers. It was designed to be introduced by the patient's provider within the existing clinic workflow, and the remainder of the intervention could be completed at home by the patient with their family.

In this aim (Aim 2), the Let's Talk cascade screening digital intervention will be pilot tested to assess feasibility for clinical use. It will be tested by genetic counselors (n=5) and their patients (n=15) who have been diagnosed with LS and are currently sharing information about their diagnosis with relatives. Genetics providers will be identified from one of three genetics clinics. After consenting to participate, they will be asked to complete a short pre-intervention survey and take part in a brief educational training to learn about the Let's Talk tool. Then, providers will help recruit eligible patients seen in one of the genetics clinics who have a need for cascade screening for Lynch Syndrome.

Once each patient enrolls, they will complete a short pre-intervention survey and then will be introduced to the online Let's Talk toolkit. They will have access to the toolkit for the following two months. The online tool was adapted from a previously developed workbook intervention guided by key stakeholders in Lynch syndrome care and patients. The toolkit addresses gaps in knowledge, self-efficacy, outcome expectancy, and other perceived barriers to cascade screening for Lynch syndrome. The adapted online tool will guide patients through the cascade screening process using evidence-based practices such as goal setting, guided practice, gain-framing, and information chunking. Patient participants will be asked to utilize the online tool to complete a variety of activities such as script writing, family tree building, and planning coping responses in the two months following enrollment.

Two months following the delivery of Let's Talk, patients will be given a brief online survey and a qualitative interview to assess outcomes (n=15). Post-intervention surveys and interviews will also be conducted with genetic counselors at the end of the study (n=5).

ELIGIBILITY:
Inclusion Criteria for Patients

* Written informed consent obtained to participate in the study.
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
* Age ≥ 18 years at the time of consent.
* Written informed consent obtained to participate in the study.
* Self-reported Lynch syndrome diagnosis.

Inclusion Criteria for Genetic Counselor

* Written informed consent obtained to participate in the study.
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
* Age ≥ 18 years at the time of consent.
* Written informed consent obtained to participate in the study.
* Self-reported employment as a practicing genetic counselor at a medical institution.

Exclusion Criteria for Patients

* The patient has already notified all relatives about their diagnosis with Lynch syndrome.

Exclusion Criteria for Genetic Counselor

* Genetic Counselor is not employed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in patient knowledge | 2 months
  Change in patient knowledge will be measured by an online survey prior to and after the intervention. Knowledge will be measured using a 12-item knowledge scale developed by Bannon et al. (2014) covering topics such as hereditary basis of Lynch syndrome (LS), transmission pattern, risks of LS-related cancers, surveillance strategies, and prophylactic options. All items on the survey are of multiple-choice format and will be scored from 0-100% based on the proportion of correct answers. Change in patient knowledge across timepoints will be analyzed using a Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Let's Talk reach | 8 months
  Reach will be calculated as the proportion of individuals who provide informed consent among those approached for participation. This proportion will be calculated based on reports from the five participating genetic counselors.
Let's Talk provider adoption | 8 months
  Adoption will be defined as the proportion of the five participating genetic providers who shared the intervention with at least one patient during the study period. This will be calculated by dividing the number of providers who report sharing the intervention with >1 patient by the total number of participating providers (n=5).
Let's Talk patient acceptability | 8 months
  Patient acceptability will be defined as patient satisfaction with the intervention. This will be evaluated using a four-item scale included in the post-intervention patient survey. Patients will indicate their level of agreement with four acceptability-related statements on a five-point Likert scale, adapted from Weiner et al. (2017), ranging from "Completely disagree" to "Completely agree".
Let's Talk provider feasibility | 8 months
  Provider feasibility will examine the extent to which providers feel they can successfully share this tool with relevant patients in a clinical setting. This will be evaluated using a four-item scale included in the end-of-study provider survey. Providers will indicate their level of agreement with four feasibility-related statements on a five-point Likert scale, adapted from Weiner et al. (2017), ranging from "Completely disagree" to "Completely agree".
Let's Talk maintenance | 8 months
  Maintenance will be defined as a provider's intention to continue sharing the Let's Talk intervention with patients after the study period ends. This will be assessed through qualitative interviews conducted at the end of each provider's participation. Providers will be asked whether they intend to continue using the tool in their practice to explain their reasoning. The proportion of providers who indicate an intention to continue using the tool will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Roberts, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials